CLINICAL TRIAL: NCT02226302
Title: Linking Obesity and Estrogen-responsive Genes in Endometrial Cancer
Acronym: FETCH
Status: Completed | Type: Observational
Sponsor: Queensland Centre for Gynaecological Cancer (Other Government)
Collaborators: Queensland Institute of Medical Research (Other); Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: FETCH
Record Dates: First submitted 2014-06-11; First posted 2014-08-27 (Estimated); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Endometrial Cancer
Keywords: Endometrial cancer; Obesity
MeSH Terms: conditions — Endometrial Neoplasms; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Omental fat samples will be stored for one year for study purposes. They will not be stored for future research
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Female Group 2: Females with BMI >30 kg/m2 who are having a hysterectomy for benign conditions
- Females Group 1: Females with BMI <30 kg/m2 who are having a hysterectomy for benign conditions
- Males: 2 males with BMI <30 kg/m2 and 2 males with BMI >30 kg/m2

SUMMARY:
The objective is to develop an organotypic model to assess the effects of obesity on the expression and methylation status of estrogen-responsive genes in endometrial cancer. Omental fat samples will be removed from participants during surgery and these fat samples will be used in laboratory analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Any patient having abdominal surgery (Laparoscopic or open technique) for benign conditions
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patients must have adequate:
* Hematologic function: Neutrophils ≥ 1.5 x 109/L and platelets ≥ 100 x 109/L
* Renal function: serum creatinine ≤ ULN or estimated glomerular filtration rate (eGFR) [CKD-EPI Formula] ≥ 60 mL/min
* Hepatic function: serum bilirubin ≤ 1.5 x ULN and AST ≤ 2.5 x ULN and ALT≤ 2.5 x ULN
* Physically able to undergo surgery
* Written informed consent

Exclusion Criteria:

* Confirmed gynaecological malignancy
* Contraindications and/or unfit for Surgery: serious concomitant systemic disorders incompatible with the study (at the discretion of the investigator);
* Patients who are pregnant or lactating
* Serious illness or medical condition but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (patients with stable AF are eligible), or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with disseminated intra-peritoneal malignancy or suspected ovarian cancer
* HIV positive
* Previous bariatric surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 12 female patients undergoing surgery for pre-existent conditions will be recruited for this study. The groups will include 6 patients with a BMI < 30 kg/m2 and 6 patients with a BMI ≥ 35 kg/m2. In addition 4 males patients will be recruited to assess responses from patients with low levels of serum estradiol.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Identify estrogen-response genes in endometrial cancer | Baseline
  Omental fat will be collected from 6 lean patients, 6 obese patients and 4 controls (male patients) and co-cultured with endometrial cancer cell lines

SECONDARY OUTCOMES:
Examine how expression of estrogen response genes are altered in obesity | Baseline
  Compare gene response in tissue from lean and obese individuals

CONTACTS AND LOCATIONS:
Overall Officials: Donal Brennan, Principal Investigator — Queensland Health
Locations (2):
- Australia (2):
  - Queen Elizabeth II Jubilee Hospital, Coopers Plains, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland